CLINICAL TRIAL: NCT02590237
Title: A Clinical Evaluation of the King Vision Video Laryngoscope aBlade System in Children
Brief Title: KingVision Video Laryngoscopy vs Direct Laryngoscopy - Equivalence Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Primary Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015-304
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Tracheal Intubation
Keywords: Laryngoscopy; Video Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Laryngoscopy (Active Comparator): The trachea will be intubated via direct laryngoscopy using a traditional straight blade (Miller) laryngoscope.
  Interventions: Device: Miller Direct Laryngoscopy
- KingVision Video Laryngoscope (Experimental): The trachea will be intubated using the Ambu KingVision Video Laryngoscope size 1 pediatric blade.
  Interventions: Device: Ambu KingVision Video Laryngoscope aBlade

INTERVENTIONS:
Device: Ambu KingVision Video Laryngoscope aBlade — At time of tracheal intubation, the subject will be intubated using the Ambu KingVision Video Laryngoscope with a size 1 aBlade. The first attempt to successful intubation will be assessed. The Cormack Lehane and Percentage of Glottic Opening scores will be recorded. Information on time to glottic view, time to removal of the blade, and time of first capnography upstroke (successful intubation) will be recorded. Other parameters measured will be information on subsequent attempts, ease of tracheal tube insertion, and hemodynamic responses for 5 minutes.
  Arms: KingVision Video Laryngoscope
Device: Miller Direct Laryngoscopy — At time of tracheal intubation, the subject will be intubated using a Miller blade laryngoscope. The first attempt to successful intubation will be assessed. The Cormack Lehane and Percentage of Glottic Opening scores will be recorded. Information on time to glottic view, time to removal of the blade, and time of first capnography upstroke (successful intubation) will be recorded. Other parameters measured will be information on subsequent attempts, ease of tracheal tube insertion, and hemodynamic responses for 5 minutes.
  Arms: Direct Laryngoscopy

SUMMARY:
The purpose of this study is to determine whether the Ambu KingVision videolaryngoscope performs as well as direct laryngoscopy for intubating small children and infants.

DETAILED DESCRIPTION:
The goal of this prospective randomized study is to compare the Ambu KingVision Video Laryngoscope and direct laryngoscopy using the Miller Blade Laryngoscope.

The primary outcome of the study will be time to successful intubation. Other outcomes of clinical relevance such as first attempt success rates of intubation, grade of laryngeal view, percentage of glottic opening, number of insertion attempts, hemodynamic responses, and complications will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Lurie Children's Hospital undergoing surgery/procedure where intubation is indicated
* American Society of Anesthesiology Class I-III patients

Exclusion Criteria:

* Children with an expected difficult airway
* A bleeding or blood clotting disorder

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Time to Intubation | Assessed intraoperatively at time of intubation
  Three timepoints will be recorded, beginning with insertion of the device past the lips into the mouth. These will include time to optimal glottic view, time to removal of device from mouth, and time to first CO2 capnography upstroke. The primary outcome measure will be total time to intubation, as the sum of all three timepoints.

SECONDARY OUTCOMES:
First Attempt Success Rate of Tracheal Intubation | Assessed intraoperatively at time of intubation
  An attempt at tracheal intubation will be defined as entry of the device into the patient's mouth without the need to remove the device once entered and securing the airway.
Grades of Laryngeal View | Assessed intraoperatively at time of intubation
  Cormack Lehane (1-4) and percentage of glottic opening (POGO) (%) will be recorded after insertion of the laryngoscope
Intubation Adjustments & Ease of Use | Assessed intraoperatively following intubation
  Airway manipulations utilized and ease of use (Likert 1-5) will be assessed by the user following the intubation.
Hemodynamic Parameters - Heart Rate | Assessed intraoperatively at time of and following intubation
  Heart rate (beats per minute) will be assessed prior to intubation and at 1 minute intervals, for 5 minutes, following intubation.
Hemodynamic Parameters - Blood Pressure | Assessed intraoperatively at time of and following intubation
  Blood pressure (mmHg) will be assessed prior to intubation and at 1 minute intervals, for 5 minutes, following intubation.
Intraoperative Complications | Assessed intraoperatively
  Airway/device related complications including, laryngospasm, bronchospasm, oxygen desaturation, will be assessed at intubation, during the surgery, and after extubation while under the anesthesiologists care.
Postoperative Complications | Assessed postoperatively while admitted to the phase 1 recovery unit, approximately 30-60 minutes after surgery
  Airway/device related complications including sore throat, hoarseness, persistent coughing, stridor, and others will be assessed in the post anesthesia care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Ann & Robert Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Levitan RM, Heitz JW, Sweeney M, Cooper RM. The complexities of tracheal intubation with direct laryngoscopy and alternative intubation devices. Ann Emerg Med. 2011 Mar;57(3):240-7. doi: 10.1016/j.annemergmed.2010.05.035. Epub 2010 Jul 31. PMID 20674088
- [Background] Theiler L, Hermann K, Schoettker P, Savoldelli G, Urwyler N, Kleine-Brueggeney M, Arheart KL, Greif R. SWIVIT--Swiss video-intubation trial evaluating video-laryngoscopes in a simulated difficult airway scenario: study protocol for a multicenter prospective randomized controlled trial in Switzerland. Trials. 2013 Apr 4;14:94. doi: 10.1186/1745-6215-14-94. PMID 23556410
- [Background] Murphy LD, Kovacs GJ, Reardon PM, Law JA. Comparison of the king vision video laryngoscope with the macintosh laryngoscope. J Emerg Med. 2014 Aug;47(2):239-46. doi: 10.1016/j.jemermed.2014.02.008. Epub 2014 Apr 16. PMID 24742495
- [Background] Akihisa Y, Maruyama K, Koyama Y, Yamada R, Ogura A, Andoh T. Comparison of intubation performance between the King Vision and Macintosh laryngoscopes in novice personnel: a randomized, crossover manikin study. J Anesth. 2014 Feb;28(1):51-7. doi: 10.1007/s00540-013-1666-9. Epub 2013 Jun 30. PMID 23812581
- [Derived] Jagannathan N, Hajduk J, Sohn L, Huang A, Sawardekar A, Albers B, Bienia S, De Oliveira GS. Randomized equivalence trial of the King Vision aBlade videolaryngoscope with the Miller direct laryngoscope for routine tracheal intubation in children <2 yr of age. Br J Anaesth. 2017 Jun 1;118(6):932-937. doi: 10.1093/bja/aex073. PMID 28549081